CLINICAL TRIAL: NCT05508529
Title: Effect of Natural Immune Modulators on Upper-Respiratory Tract Infections (URTIs) and Psychological Mood State
Brief Title: Natural Modulators of Immune Function and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3 Waves Wellness (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Immune Study 2020
Record Dates: First submitted 2022-08-13; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Stress
MeSH Terms: interventions — Nigella sativa oil; astaxanthine; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: treatment (5 dietary supplement blends) versus placebo (control)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, placebo-controlled, with coded bottles for each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Chaga Mushroom (Active Comparator): Chaga mushroom extract (1 capsule daily) Active ingredients: 480mg chaga mushroom extract Inactive ingredients: none
  Interventions: Dietary Supplement: Chaga Mushroom
- Algae Extract (Active Comparator): Algae Concentrate (2 tablets daily) Active ingredients: 8mg algae concentrate Inactive ingredients: none
  Interventions: Dietary Supplement: Algae Extract
- Black Cumin Seed Oil (Active Comparator): Black cumin seed oil (1 softgel daily) Active ingredients: 500mg black cumin seed oil Inactive ingredients: medium chain triglyceride (MCT) oil
  Interventions: Dietary Supplement: Black Cumin Seed Oil
- Black Cumin Seed Oil + Astaxanthin (Active Comparator): Black Cumin Seed Oil + Astaxanthin (3 softgels daily) Active ingredients: 500mg black cumin seed oil + 8mg astaxanthin oleoresin Inactive ingredients: medium chain triglyceride (MCT) oil
  Interventions: Dietary Supplement: Black Cumin Seed Oil + Astaxanthin
- Black Cumin Seed Oil + Omega 3 (Active Comparator): Black Cumin Seed Oil + Omega 3 (3 softgels daily) Active ingredients: 500mg black cumin seed oil + 1200mg omega3 from 1500mg fish oil Inactive ingredients: none
  Interventions: Dietary Supplement: Black Cumin Seed Oil + Omega 3
- Placebo (Placebo Comparator): Placebo (1 capsule daily) Inactive ingredients: 500 mg Cornstarch/Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chaga Mushroom — Effect of chaga on immune/mood support
  Arms: Chaga Mushroom
Dietary Supplement: Algae Extract — Effect of algae extract on immune/mood support
  Arms: Algae Extract
Dietary Supplement: Black Cumin Seed Oil — Effect of black cumin seed oil on immune/mood support
  Arms: Black Cumin Seed Oil
Dietary Supplement: Black Cumin Seed Oil + Astaxanthin — Effect of Black Cumin Seed Oil + Astaxanthin blend on immune/mood support
  Arms: Black Cumin Seed Oil + Astaxanthin
Dietary Supplement: Black Cumin Seed Oil + Omega 3 — Effect of Black Cumin Seed Oil + Omega3 blend on immune/mood support
  Arms: Black Cumin Seed Oil + Omega 3
Dietary Supplement: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The objective of this proposal is to recruit 20 healthy subjects per ingredient arm (5 arms x 20 subjects; N= 120 total) to participate in a research study investigating the effects of dietary supplementation for one-month with different dietary supplement formulations (versus placebo; N=20) that may have benefits for supporting respiratory health, psychological stress, and quality of life.

Supplements to be studied (all are commercially available):

1. Chaga (mushroom extract)
2. Arava (algae concentrate)
3. Thymoquin (black cumin seed oil)
4. Thymoquin + Astaxanthin (antioxidant carotenoid)
5. Thymoquin + Omega 3 (fish oil)
6. Placebo (corn starch)

In order to "stress" volunteers, participants will train for and complete a strenuous off-road trail marathon to induce both physical and mental stress.

DETAILED DESCRIPTION:
The main hypothesis is that the group(s) supplementing with natural stress modulators will demonstrate superior subjective assessments of both physical health (e.g. respiratory function, mobility, flexibility) and mental stress (e.g. mood, energy, focus).

Stress-related factors following intense endurance activity can lead to a range of adverse physical manifestations including muscle soreness, physical fatigue, and general malaise. Furthermore, stressful events frequently lead to negative emotions including temporary reductions in perceived mood and energy with heightened irritability and tension.

Each of the ingredients under consideration for this study, Chaga, Algae extract, Black Cumin Seed Oil, Astaxanthin, and Omega-3s, have a number of laboratory and animal studies demonstrating anti-stress benefits including improvements in physical mobility (e.g. flexibility), mental energy, and overall well-being.

Each of these ingredients may be considered as natural "stress-modulators" that can help to balance overall well-being and quality of life. Such natural substances represent an emerging approach to buffer the detreimnetal effects of physical and mental stressors.

Mushrooms, particularly Chaga, have a long history of use in traditional medicine for supporting general well-being. An abundance of in-vitro evidence suggests that a wide range of mushroom bioactives may modify stress responses, with promising preliminary research in humans.

Algae concentrate and in particular Astaxanthin, the natural red carotenoid pigment found in microalgae, has been shown to be a broad-spectrum stress modulator, likely due to its actions in reducing oxidative and inflammatory stress and thus protecting mitochondria from damage and controlling cellular senescence.

Black cumin seed oil and its primary bioactive compound, thymoquinone, have been used in traditional Middle Eastern Medicine for thousands of years for its broad-spectrum benefits related to longevity and overall well-being.

Omega-3 fatty acids are well-described in the scientific literature for their anti-inflammatory effects and thus benefits in a wide range of health parameters. Because of the close relationship between well-being and inflammatory balance, omega-3 fatty acids may help to support quality of life parameters, particularly after stress, which is known to disrupt both inflammatory signaling and psychological mood state.

Key Outcome Measures

* Mental and Physical Stress (Vivosmart)
* Mood, Energy, Focus, etc = Profile of Mood States (POMS)
* Microbiome Assessment (BiomeTracker)
* Salivary Cortisol (morning waking sample)
* Well-Being Symptoms (Health Log)
* Blood Pressure (in 4 arms containing Black Cumin Seed OIl and Placebo)
* Blood Omega 3 (in 2 arms containing Omega3 and Placebo)

Volunteers will perform all study measurements in the privacy of their own home.

Mental & Physical Stress

* Stress (mental and physical) is assessed by heart rate variability (the time interval between heart beats)
* "Readiness" is assessed as "Body Battery Energy" - a combination assessment of stress, heart rate variability, sleep quality, and physical activity.
* Sleep Quality is assessed by tracking total, light, deep, and REM stages of sleep.
* Each of these parameters is automatically uploaded by the subject to a secure password-protected online database (Garmin Connect) where the investigators can access to collect and collate data.

Health Log The daily health log contains questions related to overall health status and general well-being (e.g. stress, energy, flexibility/mobility, etc).

Mood Assessment (POMS; Profile of Mood States) Longer term changes in mood/focus/energy will be assessed using the research-validated Profile of Mood States (POMS) questionnaire to measure 6 primary psychological factors (tension, depression, anger, fatigue, vigor, or confusion) plus the combined global mood state as an indication of subjective well-being. The POMS methodology has been used in ~3,000 studies, and its validity is well established. The POMS profile uses 65 adjective-based intensity scales scored on a 0-4 hedonic scale (e.g. "not at all" to "extremely"). The 65 adjective responses are categorized into the 6 mood factors (tension, depression, anger, fatigue, vigor, or confusion), tabulated, scored, and analyzed. The output of the POMS questionnaire is an assessment of the positive and negative moods of each subject at baseline and post-supplementation.

Microbiome Assessment (BiomeTracker) Microbiome analysis of fecal samples will be carried out using the complete BiomeTracker system (Wasatch Scientific, Murray, UT). Briefly, fecal samples will obtained by nylon swab and placed into preservative binding buffer to lock the composition of bacteria in place. DNA is then purified using DNA columns and ~20ng of DNA from each sample is added to the reaction mixtures. Samples are processed on an ABI 7500 Fast (Applied Biosystems) instrument in duplicate. A "microbiome composite score" is generated as an overall average of many different aspects of microbiome balance, including Bifidobacterium, Lactobacillus, Akkermansia, Firmicutes/Bacteroidetes (F/B) ratio, and others.

Volunteers will be provided with take-home kit to obtain fecal samples in the privacy of their home for analysis. The kit will include detailed instructions and postage paid packaging to be returned directly to Wasatch Scientific Laboratories. Each kit will be numerically coded so that samples are blinded to the lab.

Salivary Cortisol Cortisol is the major glucocorticosteroid hormone produced in the adrenal cortex. Cortisol is actively involved in the regulation of calcium absorption, blood pressure maintenance, anti-inflammatory function, gluconeogenesis, gastric acid, pepsin secretion, and immune function. Cortisol production has a circadian rhythm. Levels peak in the early morning and drop to the lowest concentration at night. Levels rise independently of circadian rhythm in response to stress. In the blood only 1 to 15% of cortisol is in its unbound or biologically active form. The remaining cortisol is bound to serum proteins. Unbound serum cortisol enters the saliva via intracellular mechanisms, and in saliva the majority of cortisol remains unbound to protein. Salivary cortisol levels are unaffected by salivary flow rate or salivary enzymes. Studies consistently report high correlations between serum and saliva cortisol, indicating that salivary cortisol levels reliably estimate serum cortisol levels.

Volunteers will be provided with take-home kit to obtain saliva samples in the privacy of their home for cortisol analysis. The kit will include detailed instructions and will be returned to CRC for shipment to Wasatch Scientific Laboratories. Each kit will be numerically coded so that samples are blinded to the lab.

The CRC will confirm with volunteers and Wasatch Scientific that these samples have been collected and received by the lab for analysis.

Blood Pressure Blood pressure will be measured with Omron Series 3 Upper Arm Blood Pressure Monitor, which will be provided to 10 randomly selected participants in each of the three study arms containing Thymoquin as well as 10 randomly selected participants in the placebo group.

Blood Omega-3 Index Blood levels of omega-3 fatty acids will be assessed in the group taking Omega-3 fish oil supplements, using a self-collected at-home fingerstick blood sample (OmegaQuant). Subjects will receive all supplies and instructions (see Instruction card below) to apply a drop of blood to the collection card and mail sample to the laboratory in a pre-paid envelope.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18 to 60 years
* Ability to complete strenuous off-road trail run, and planning to do so regardless of the study
* Willingness to consume the dietary supplements under investigation
* Willingness to undertake all protocol measurements and training regimens
* Ability to understand and sign the informed consent form (ICF)

Exclusion Criteria:

* Any supplements or medications that are stress/immune-suppressive or stress/immune-stimulant (e.g. herbal stimulants).
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Psychological Mood State (e.g. stress) | 1 month
  "Global Well-Being" index as collected by the validated Profile of Mood States Survey (POMS)
Health Log | 1 month
  total number of subjective upper respiratory tract complaints per subject (e.g. sore throat, cough, etc)
Stress Hormones | 1 month
  Salivary Cortisol (ng/ml)
Microbiome Balance | 1 month
  Streptococcus thermophilus (relative abundance)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Talbott, PhD, Principal Investigator — 3 Waves Wellness
Locations (1):
- 3 Waves Wellness, LLC, Plymouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon study completion
Access Criteria: data will be available upon request

REFERENCES:
- [Background] Talbott SM, Talbott JA, Talbott TL, Dingler E. beta-Glucan supplementation, allergy symptoms, and quality of life in self-described ragweed allergy sufferers. Food Sci Nutr. 2013 Jan;1(1):90-101. doi: 10.1002/fsn3.11. Epub 2014 Jan 8. PMID 24804018
- [Background] Talbott SM, Talbott JA, George A, Pugh M. Effect of Tongkat Ali on stress hormones and psychological mood state in moderately stressed subjects. J Int Soc Sports Nutr. 2013 May 26;10(1):28. doi: 10.1186/1550-2783-10-28. PMID 23705671
- [Background] Talbott SM, Talbott JA. Baker's yeast beta-glucan supplement reduces upper respiratory symptoms and improves mood state in stressed women. J Am Coll Nutr. 2012 Aug;31(4):295-300. doi: 10.1080/07315724.2012.10720441. PMID 23378458
- [Background] Talbott SM, Talbott JA, Pugh M. Effect of Magnolia officinalis and Phellodendron amurense (Relora(R)) on cortisol and psychological mood state in moderately stressed subjects. J Int Soc Sports Nutr. 2013 Aug 7;10(1):37. doi: 10.1186/1550-2783-10-37. PMID 23924268